CLINICAL TRIAL: NCT01910493
Title: Evaluation of the Impact of Mobile Phone Messages on ART and PMTCT Adherence in Mozambique: A Randomized Control Trial
Brief Title: Evaluation of the Impact of Mobile Phone Messages on ART and PMTCT Adherence in Mozambique
Acronym: SMSaude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Absolute Return for Kids (Other)
Collaborators: Vodacom (Unknown); United States Agency for International Development (USAID) (U.S. Federal Agency); Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMSaude01
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV-positive
Keywords: mhealth; mobile health; SMS; SMS reminders; ART retention in care; PMTCT; PMTCT cascade; retention in care
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ART no SMS reminders (Active Comparator): control group
  Interventions: Behavioral: SMS reminders
- PMTCT no SMS reminders (Active Comparator): control group
  Interventions: Behavioral: SMS reminders
- SMS reminders to PMTCT cohort (Experimental): experimental group
  Interventions: Behavioral: SMS reminders
- SMS reminders to ART cohort (Experimental): experimental group
  Interventions: Behavioral: SMS reminders

INTERVENTIONS:
Behavioral: SMS reminders — Intervention participants only will be sent text messages to their phones. The content of text messages will have a maximum of 160 characters and not mention HIV and will state the dates for the forthcoming consultations, visits to the pharmacy, lab results, time to take medication and reminders for patients who miss appointments.

SUMMARY:
Mobile phone SMS are increasingly used to promote positive health behaviour with an aim to improve health outcomes. However, robust data on the efficacy of SMS on health seeking behaviour and patient outcomes in resource-limited settings is sparse. The SMSaude study aims to assess whether regular SMS-reminders improve retention on antiretroviral therapy (ART) and prevention of mother to child transmission of HIV (PMTCT) programmes in Mozambique.

DETAILED DESCRIPTION:
SMSaúde is a multisite randomised clinical trial of HIV-infected adults on ART and HIV-infected pregnant women in six clinics in Maputo Province, Mozambique. Eligibility criteria include: currently residing in the province; no plans to move for 12+ months; have own cell-phone; literate; 8-28 weeks pregnant (PMTCT cohort); on first line ART and on ART for >15 days (ART cohort). Patients were interviewed for eligibility, and then randomized (1:1). SMS reminders are sent to the intervention group using software that picks up the patient's next appointment from the electronic patient database. Primary outcomes tested were improved retention in ART care and uptake of all PMTCT services.

ELIGIBILITY:
Inclusion Criteria:

* On ART for >15 days (for ART only)
* Live in province and plan to stay for 12+ months
* Have cell phone
* Literate

For PMTCT (in addition to above criteria):

- pregnant between 8-28 weeks

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1352 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Retention in ART care | 12 months

SECONDARY OUTCOMES:
Retention in PMTCT care | until 8 weeks post partum

CONTACTS AND LOCATIONS:
Overall Officials: Cesar de Palha, MD, Principal Investigator — University of Eduardo Mondlane
Locations (1):
- 6 Health Facilities, Matola, Xinavane, Machava and Namaacha, Maputo, Mozambique